CLINICAL TRIAL: NCT05115019
Title: A Phase II/III, Double-blind, Randomized, Placebo-controlled Clinical Trial to Evaluate the Efficacy of RUTI® to Reduce the Severity of SARS-CoV-2 Infection
Brief Title: A Clinical Trial to Evaluate the Efficacy of RUTI® to Reduce the Severity of SARS-CoV-2 Infection (COVID-19)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decrease of incidence and severity of COVID and availability of therapeutic alternatives
Sponsor: PT. Innovative Pharma Solutions (Industry)
Collaborators: Archivel Farma S.L. (Industry); RUTI Immunotherapeutics S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYCOVIND
Record Dates: First submitted 2021-11-09; First posted 2021-11-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (RUTI) (Experimental): Participants will receive one dose of RUTI® vaccine at the baseline visit, which will be administered subcutaneously in the deltoid region at a dose of 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli (FCMtb) in an injection volume of 0.3 m
  Interventions: Biological: RUTI® vaccine
- Group B (Placebo) (Placebo Comparator): Participants will receive one dose of sterile physiological serum at the baseline visit, which will be administered subcutaneously in the deltoid region.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® vaccine — Each dose of the RUTI® vaccine contains 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli (FCMtb) in a total volum of 0.3mL.
  Arms: Group A (RUTI)
Biological: Placebo — Physiological serum, 0.9% NaCl, will be used as a placebo
  Arms: Group B (Placebo)

SUMMARY:
The aim of this study is to assess the efficacy of the RUTI® vaccine in achieving clinical improvement of COVID-19 symptoms and to evaluate the safety of RUTI® in patients with SARS-CoV-2 infection. The study will include a comparison between placebo and RUTI® vaccine in a 1:1 design.

DETAILED DESCRIPTION:
Once it has been confirmed that the patient meets the selection criteria, subjects will be randomly assigned to one of the two study groups:

* Experimental group: Administration of RUTI®
* Control group: Administration of Placebo (physiological serum)

This randomization follows a 1:1 ratio. In this way, of the total of 550 subjects who intend to be recruited for this study, 275 will receive the prophylactic treatment, and 275 will receive the placebo treatment.

Neither patient nor the doctor will know if the subject is part of the experimental group or the control group, that is to say, the treatment assignment is blind.

All subjets will receive just one inoculation of treatment (either RUTI® or Pacebo). The standard treatment of COVID-19, if is necessary, will continue after RUTI® administration according to the local guidelines.

All the subjets will be followed for one month after the first day of RUTI® or Placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent before initiating the selection procedures.
2. Patients infected with SARS-CoV-2 (PCR +) with mild symptoms up to 7 days that do not require hospitalization, from the onset of symptoms. Mild symptoms, defined as the following criteria: cough, headache, fever (>37.5ºC), muscular pain and shortness of breath.
3. People ≥ 18 years.
4. Peripheral oxygen saturation (SpO2) more than 94% on room air, not requiring supplemental oxygen.
5. Availability to meet the requirements of the protocol.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Suspected of active viral or bacterial infection other than SARS-CoV-2.
3. Participation in another interventional study with potentially conflicting medication within 30 days before screening.
4. Severely immunocompromised people (data gathered from preexisting medical records and history taking). This exclusion category includes:

   1. Subjects with human immunodeficiency virus (HIV-1).
   2. Neutropenic subjects with less than 500 neutrophils / mm3.
   3. Subjects with solid organ transplantation.
   4. Subjects with bone marrow transplantation.
   5. Subjects undergoing chemotherapy.
   6. Subjects with primary immunodeficiency.
   7. Severe lymphopenia with less than 400 lymphocytes / mm3.
   8. Treatment with any anti-cytokine therapy.
   9. Oral treatment with steroids, defined as daily doses of 10 mg prednisone or equivalent for more than 3 months.
5. Malignancy, or active solid or non-solid lymphoma from the previous two years.
6. BCG vaccination in the last 10 years.
7. Chloroquine or hydroxychloroquine administration in the last two weeks
8. Soy allergy
9. Direct involvement in the design or execution of the MYCOVIND clinical trial.
10. Do not have a smartphone.
11. Detection by the investigator of lack of knowledge or willingness to participate and comply with all requirements of the protocol.
12. Any other findings that, at the discretion of the investigator, may compromise compliance with the protocol or that may influence significantly the interpretation or the results of the effects of probiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Reduction patient rate to category 0 according to the WHO Ordinal scale by Day 30 after the initiation of vaccination | 1 month
  Reduction patient rate to category 0 according to the WHO Ordinal scale by Day 30 after the initiation of vaccination

SECONDARY OUTCOMES:
Fever | 1 month
  Number of days with fever (≥38 ºC).
Incidence of acute respiratory symptoms | 1 month
  Number of acute respiratory symptoms (SpO2 < 95%)
Patient rate reduction C1 or lower (WHO scale) | 1 month
  Reduction patient rate to category 1 or lower according to the WHO Ordinal scale
Incidence of death by SARS-CoV | 1 month
  Accumulated Incidence of death by SARS-CoV
Incidence admission at Intensive Care Unit | 1 month
  Accumulated incidence admission at Intensive Care Unit (documented)
Days in Intensive Care Unit | 1 month
  Number of days in Intensive Care Unit (documented)
Incidence for mechanic ventilation due to SARS-CoV-2 infection | 1 month
  Accumulated incidence for mechanic ventilation due to SARS-CoV-2 infection (documented)
Days of mechanic ventilation due to SARS-CoV-2 infection | 1 month
  Number of days of mechanic ventilation due to SARS-CoV-2 infection
Days hospital admission due to SARS-CoV-2 infection | 1 month
  Number of days hospital admission due to SARS-CoV-2 infection
Incidence of Treatment-Emergent Adverse Events | 1 month
  Proportion of patients reporting Adverse events (AEs, including serious adverse events)
Levels of IgG SARS-CoV2 | 1 month
  Plasma SARS-CoV2 spike protein-specific IgG level